CLINICAL TRIAL: NCT03441750
Title: A Multicentre, Open-labelled, Randomized, Controlled Study to Evaluate the Efficacy of Metformin in Preventing Diabetes in China.
Brief Title: Efficacy of Metformin in Preventing Diabetes in China
Acronym: ChinaDPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese Association of Geriatric Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ChineseAGR
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- metformin plus standard lifestyle intervention (Experimental): Metformin starting dose is 850mg/d, it will be titrated to 850mg twice daily after 2 weeks and maintained until the last subject completes 2 years' intervention.
  Interventions: Drug: metformin
- Standard lifestyle intervention (Other): Standard lifestyle advice will be united for all subjects by providing special booklet.
  Interventions: Other: Standard lifestyle intervention

INTERVENTIONS:
Drug: metformin — Metformin tablets will be administrated in the experimental arm.
  Other Names: Glucophage immediate release formulation
  Arms: metformin plus standard lifestyle intervention
Other: Standard lifestyle intervention — Standard lifestyle advice will be united for all subjects by providing special booklet.
  * All participants will receive 20-30 minutes individual or group session with assigned nurse addressing the harm of prediabetes and the importance of a healthy lifestyle for preventing Diabetes.
  * The amount of energy intake of the participants will be calculated based on the ideal body weight and physical activity levels. The sample recipe will be explained by the nurse and provided in the diet instruction.
  * Moderate intensity physical activity (150 minutes per week) is recommended.
  * Smoking cessation is encouraged for the smoker.
  * Excessive alcohol intake is encouraged to avoid.
  Arms: Standard lifestyle intervention

SUMMARY:
A multicentred, randomized, open study to evaluate the efficacy of metformin in preventing Diabetes.

DETAILED DESCRIPTION:
The increasing prevalence of prediabetes had been documented in the recent national surveillance in China. Prediabetes is an important risk factor for developing overt Diabetes and macro/micro vascular diseases. Pharmaceutical medications such as metformin had been proved effective in preventing Diabetes. Local studies are in need to guide the clinicians in their daily practice to prevent Diabetes in China. Therefore, China Diabetes Prevention Program（China DPP）is designed and conducted to compare the efficacy of metformin combined with lifestyle intervention versus lifestyle intervention alone in preventing Diabetes.

ELIGIBILITY:
Main Inclusion Criteria:

1. Diagnosis of IGR before the randomization based on the 1999 WHO diagnostic and classification criteria.
2. Age: 18 ≤age≤70 years old.
3. Not on a treatment of anti-diabetic agents, including Chinese traditional herbs lowering blood glucose for at least 6 months before screening.
4. Male or non-pregnant, non-breastfeeding females, females without birthing plan in next three years.
5. Body mass index (BMI) ：21 kg/m2 ≤BMI<32 kg/m2.
6. Written informed consent given before any trial-related activities are carried out.

Main exclusion Criteria:

1. Administration with medications for pre-existed diseases affect glucose metabolism (except thiazide diuretics when its daily dose≤12.5mg).
2. Administration with anti-obesity agents (including Chinese traditional medicine) within 6 months of enrolment and during intervention.
3. Administration with three or more than three types antihypertensive drugs.
4. Diabetes patients (subjects with prior history of gestational Diabetes will not be excluded).
5. Have any of the following cardiovascular conditions within 3 months prior to the screening visit: acute myocardial infarction, congestive heart failure defined as New York Heart Association class III/IV or left ventricular ejection fraction ≤40%,) or cerebrovascular accident.
6. Persistent uncontrolled hypertension (systolic blood pressure ≥160mmHg, or diastolic blood pressure ≥100 mmHg).
7. Impaired liver function, have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, ALT or AST levels ≥3 times the upper limit of the reference range at the screening visit.
8. Renal dysfunction (eGFR<45ml/min）.
9. Patients ventilated by ventilator.
10. Hypersensitivity to metformin or to any of the excipients such as povidone K 30, magnesium stearate and hypromellose.
11. Disease which may cause tissue hypoxia (especially acute disease, or worsening of chronic respiratory disease).
12. Acute alcohol intoxication, alcoholism.
13. Severe chronic gastrointestinal disease.
14. Severe psychiatric illness.
15. Cancer requiring treatment in past 5 years.
16. Uncontrolled thyroid diseases.
17. Women who are pregnant or breastfeeding .
18. Participation in another clinical trial within the past 30 days .
19. Other significant disease that in the Investigator's opinion would exclude the subject from the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1724 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of newly diagnosed diabetes | The primary outcome will be evaluated when the last subject completes 2 years' intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Guangwei Li, M.D., Ph.D., Principal Investigator — Chinese Association of Geriatric Research
Locations (1):
- The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang L, Zhang Y, Shen S, Wang X, Dong L, Li Q, Ren W, Li Y, Bai J, Gong Q, Kuang H, Qi L, Lu Q, Cheng W, Liu Y, Yan S, Wu D, Fang H, Hou F, Wang Y, Yang Z, Lian X, Du J, Sun N, Ji L, Li G; China Diabetes Prevention Program Study Group. Safety and effectiveness of metformin plus lifestyle intervention compared with lifestyle intervention alone in preventing progression to diabetes in a Chinese population with impaired glucose regulation: a multicentre, open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2023 Aug;11(8):567-577. doi: 10.1016/S2213-8587(23)00132-8. Epub 2023 Jul 3. PMID 37414069
- [Derived] Ji L, Sun N, Zhang Y, Zhang L, Shen S, Wang X, Li Q, Dong L, Ren W, Qi L, Li Y, Yan S, Cheng W, Kuang H, Li G. Efficacy of metformin in preventing progression to diabetes in a Chinese population with impaired glucose regulation: Protocol for a multicentre, open-label, randomized controlled clinical study. Diabetes Obes Metab. 2020 Feb;22(2):158-166. doi: 10.1111/dom.13884. Epub 2019 Oct 24. PMID 31512365